CLINICAL TRIAL: NCT07033390
Title: Adaptation of Monitor Orthopaedic Footwear Questionnaire (MOS) Into Turkish: Validity and Reliability Study
Brief Title: Monitor Orthopaedic Footwear Questionnaire (MOS) Validity and Reliability Study
Acronym: MOS
Status: Enrolling by invitation | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Hande YAZICI, Lecturer, Medipol University
Other Study IDs: İsciH
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Validity and Safety
Keywords: validity; reability; orthopedic shoes; survey
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey — validity and reliability study of MOS

SUMMARY:
The aim of the study is to adapt the MOS questionnaire into Turkish and to investigate the validity and reliability of the questionnaire. In this study, Monitor Orthopaedic Shoes Questionnaire (MOS) will be translated into Turkish and named as MOS-T.

The research is a methodological study conducted to determine the validity and reliability of the Turkish adaptation of the MOS. For this purpose, the questionnaire will be translated into Turkish, cultural adaptation of the Turkish version will be made, and its validity and reliability will be tested.In accordance with the validity and reliability research, MOS will be reapplied to the participants after 8 weeks to evaluate the test-retest reliability.

Inclusion Criteria

* Wearing orthopaedic shoes for the first time,
* 16 years of age or older,
* Native language is Turkish and at least literacy level,
* Able to complete the questionnaire without assistance with cognitive or physical impairments,
* Who volunteered to participate in the study

DETAILED DESCRIPTION:
The translation procedure and cross-cultural adaptation of the MOS will be carried out according to the predetermined cross-cultural adaptation principles of Beaton et al. For the development of the Turkish adaptation of the MOS and the validity and reliability study, permission was obtained by e-mail from Jaap Van Netten, the first author of the original questionnaire. Firstly, two independent translators will translate the original questionnaire from English to Turkish. One of the translators will be informed about the study, the other will not be informed about the study. A draft version, which is a synthesis of these two different translations, will be prepared by a team of experts from different disciplines. The draft version will be back-translated from Turkish to English by two independent translators who are native speakers of English and fluent in Turkish to ensure that the translation expresses the same article content as the original English version. The expert team will review the translated English version and finalise the Turkish draft by deciding whether the Turkish version reflects the content of the original MOS. Finally, a pilot study will be conducted to test the items to be modified and deleted before the final Turkish version is created. After the pilot study, the final version of the Turkish version of the MOS will be created.

ELIGIBILITY:
Inclusion Criteria:

* • Wearing orthopedic shoes for the first time,

  * Being 16 years old and above,
  * Being a native Turkish speaker and having at least a literacy level,
  * Being able to complete the survey without assistance regarding cognitive or physical disorders,
  * Volunteering to participate in the study

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals using insoles
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
validity | 2-month change
  RMSEA and CFI values in confirmatory factor analysis
reliability | 2-month change
  Cronbach's alpha and ICC value

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Beykoz, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided